CLINICAL TRIAL: NCT00725959
Title: Online Social Networking for HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado School of Public Health (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Internet Sexuality Information Services (ISIS) (Other); Columbia University (Other); Rutgers University (Other)
Responsible Party: Principal Investigator, Sheana Bull, Professor, Colorado School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMIRB 07-0459; R01NR010492 (NIH); 1R01NR01492-01
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: HIV Prevention; Social Networking; Technology Based Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Facebook Arm (Experimental): Participants in this arm will have exposure to innovative, dynamic and regularly updated HIV Prevention messages on Facebook
  Interventions: Behavioral: Online social networking HIV prevention
- Control arm (Active Comparator): Participants in this arm will have exposure to static information on HIV prevention currently available online
  Interventions: Behavioral: Online social networking HIV prevention

INTERVENTIONS:
Behavioral: Online social networking HIV prevention — messages about HIV posted in online social networking sites

SUMMARY:
In this randomized controlled trial, we will identify social networks on Facebook, an randomly assign each network to control or intervention status. We will then intervene at the level of the network with dynamic, interactive HIV prevention messages (intervention) or static messages about HIV prevention (control). We will develop the intervention content with input from our target audience (Facebook users) and will measure baseline, and 3 and 6 month assessments of condom use and abstinence among all participants

ELIGIBILITY:
Inclusion Criteria:

* Facebook user with an existing Facebook page
* at least 16
* no older than 24
* English speaker

Exclusion Criteria:

* older than 24 or younger than 16
* non English speaker
* does not have a Facebook page

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1578 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheana Bull, Ph.D., Principal Investigator — University of Colorado at Denver and Health Sciences

REFERENCES:
- [Derived] Bull SS, Levine DK, Black SR, Schmiege SJ, Santelli J. Social media-delivered sexual health intervention: a cluster randomized controlled trial. Am J Prev Med. 2012 Nov;43(5):467-74. doi: 10.1016/j.amepre.2012.07.022. PMID 23079168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began October 2010 and Ended May 2011 in community settings
Groups:
- Intervention Arm: Group exposed to dynamic content on Facebook re: HIV Prevention
- Control Arm: Attention Control exposed to a current events Facebook page
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 942 | 636
Completed | 653 | 439
Not Completed | 289 | 197

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Group exposed to dynamic content on Facebook re: HIV Prevention
- Arm 2: Attention Control exposed to a current events Facebook page
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 942 | 636 | 1578
Age, Continuous [Mean (Standard Deviation); unit: years] — Years of age
  years | 19.7 (2.0) | 20.2 (2.4) | 19.8 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521 | 391 | 912
  Male | 421 | 245 | 666

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Condom Usage
Description: number of times condom used divided by number of times person had sex in past 60 days
Time Frame: two months
Measure: Mean (95% Confidence Interval); unit: proportion of condom use
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 653 | 439
proportion of condom use | .68 [.56 to .74] | .56 [.48 to .61]

2. Secondary Outcome: Condom and Abstinence Norms, Attitudes, Self-efficacy and Intentions
Time Frame: two months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: throughout entire enrollment and study follow up periods
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/942 | 0/636
Serious Adverse Events (participants affected / at risk) | 0/942 | 0/636
Other Adverse Events (participants affected / at risk) | 0/942 | 0/636

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No